CLINICAL TRIAL: NCT01090700
Title: A Phase I, Open-label, Randomized, 3-way Crossover Trial in Healthy Subjects to Investigate the Pharmacokinetic Interaction Between TMC435 and Escitalopram at Steady-state
Brief Title: TMC435-TiDP16-C112 - Interaction Trial With Antidepressants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR017044
Record Dates: First submitted 2010-03-11; First posted 2010-03-22 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Hepatitis C Virus
Keywords: TMC435-TiDP16-C112; TMC435-C112; TMC435; HCV; Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir; Escitalopram

ARMS (3):
- 001 (Experimental): TMC435 TMC435 150 mg daily for 7 days
  Interventions: Drug: TMC435
- 002 (Other): Escitalopram Escitalopram 10 mg daily for 7 days
  Interventions: Drug: Escitalopram
- 003 (Experimental): TMC435 + Escitalopram TMC435 150 mg + escitalopram 10 mg daily for 7 days
  Interventions: Drug: TMC435 + Escitalopram

INTERVENTIONS:
Drug: TMC435 — TMC435 150 mg daily for 7 days
  Arms: 001
Drug: Escitalopram — Escitalopram 10 mg daily for 7 days
  Arms: 002
Drug: TMC435 + Escitalopram — TMC435 150 mg + escitalopram 10 mg daily for 7 days
  Arms: 003

SUMMARY:
The purpose of this study is to investigate the effect of steady-state concentrations of TMC435 150mg q.d. (once a day) on the steady-state pharmacokinetics of escitalopram 10 mg q.d., and vice versa. Steady state is a term which means that the drug has been given long enough so that the plasma concentrations will remain the same with each subsequent dose. TMC435 is being investigated for the treatment of chronic hepatitis C virus (HCV) infection. Pharmacokinetics (pk) means how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body.

DETAILED DESCRIPTION:
TMC435 is being investigated for treatment of chronic HCV infection, in combination with Peg-IFN (pegylated interferon) and RBV (ribavirin). Peg-IFN plus RBV are currently an accepted methods for treating HCV. Treatment with Peg-IFN plus RBV for HCV infection is associated with a high rate of depression. The results of this study will provide dosing recommendations for coadministration of TMC435 and escitalopram in HCV-infected patients. This is a Phase I, open-label (both participant and investigator know the name of the medication) , randomized (study medication assigned by chance), crossover trial in 18 healthy participants to investigate the pharmacokinetic interaction between escitalopram and TMC435, both at steady state. Steady state is a term which means that the drug has been given long enough so that the plasma concentrations will remain the same with each subsequent dose. The participants will receive three treatments (treatment A-B-C) in a randomized order. In Treatment A, participants will receive TMC435 150 mg q.d. In Treatment B, participants will receive escitalopram 10 mg q.d. In treatment C, participants will receive escitalopram 10 mg q.d. and TMC435 150 mg q.d. All treatments will be administered for 7 days and with food. There will be a washout period (a period where no treatment will be taken in view of having all the medication eliminated from the body before starting a new treatment) of at least 10 days between last intake of study medication in one session and first intake of study medication in the subsequent session. Pharmacokinetic profiles of the two compounds will be measured through blood samples taken at regular intervals during the study and safety and tolerability will be assessed during the study period and in follow-up. Safety and tolerability evaluations will be recorded at regular intervals throughout the trial period. Blood and urine samples, electrocardiogram (ECG) and vital signs (blood pressure and heart rate) will be taken at screening, before medication intake on days 1 and 7 and on Day 8 in each session and at the 2 follow up visits at 1 week and 4-5 weeks after last dose of drug in the last session. A physical examination will be performed at screening, on day -1 (= day before day of first medication intake in each session) and during the 2 follow up visits. On the morning before first medication intake (in the first session only) a blood sample will be taken to examine your CYP2C19 genes, which are responsible for the production of enzymes that determine the breakdown of drugs in your body. The results of this study will provide dosing recommendations for coadministration of TMC435 and escitalopram in HCV-infected patients. Participants will receive in treatment A TMC435 150 mg q.d., in treatment B participants will receive escitalopram 10 mg and in treatment C participants will receive escitalopram 10 mg q.d. + TMC435 150 mg q.d. All treatments will be administered for 7 days and with food.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers for at least 3 months prior to screening
* Healthy on the basis of physical examination, medical history, vital signs and 12-lead ECG performed at screening
* Healthy on the basis of clinical laboratory tests performed at screening
* Subjects must have signed an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study
* Participants must have signed the ICF for pharmacogenetic research indicating willingness to participate in the pharmacogenetic component of the study.

Exclusion Criteria:

* A positive human immunodeficiency virus - type 1 (HIV-1) or HIV-2 test at study screening
* Hepatitis A, B, or C infection (confirmed by hepatitis A antibody immunoglobulin [IgM], hepatitis B surface antigen, or hepatitis C virus antibody, respectively) at screening
* History of liver or renal (estimated creatinine clearance below 60 mL/min) insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal (such as significant diarrhea, gastric stasis, or constipation that in the investigator's opinion could influence drug absorption or bioavailability), endocrine, neurologic, hematologic, rheumatologic, psychiatric and neoplastic or metabolic disturbances
* Known allergies, hypersensitivity, or intolerance to TMC435 or its excipients
* Received an investigational drug (including investigational vaccines) or used an investigational medical device within 60 days before the planned start of treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of stable blood levels of TMC 435 given 150 mg q.d. on the stable blood levels of escitalopram given 10 mg q.d. in healthy participants and vica versa. | pk profiles of TMC435 will be measured up to 24 hours on Day 7 in Treatment A and C. Pharmacokinetic profiles of escitalopram will be measured up to 24 hours postdose on Day 7 of Treatment B and C.

SECONDARY OUTCOMES:
The short-term safety and tolerability of coadministration of TMC435 and escitalopram in healthy participants (safety and tolerability criteria are the activity of the heart, blood pressure, pulse, physical examination, parameters in urine and blood) | This will be determined throughout the study; Day-1 through Day 8 in each session, 1 week and 4-5 weeks after last medication intake

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited